CLINICAL TRIAL: NCT01109927
Title: Early Insulin Treatment in Patients With Latent Autoimmune Diabetes (LADA)
Brief Title: Early Insulin Treatment in Patients With Latent Autoimmune Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lund University Hospital (Other)
Collaborators: Landstinget Kronoberg, Sweden (Unknown)
Responsible Party: Mona Landin-Olsson, prof, Dept of Clinical Science, Lund University Hospital, Lund, Sweden, Lund University Hospital, Lund, Sweden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LundUH-LADA101
Record Dates: First submitted 2010-04-08; First posted 2010-04-23 (Estimated); Last update posted 2010-04-23 (Estimated); Status verified 1995-02

CONDITIONS: Diabetes, Autoimmune; Diabetes Mellitus, Adult-Onset
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin treatment (Experimental): Insulin given as soon as possible after diagnosis
  Interventions: Drug: Insulin
- Conventional treatment (No Intervention): Diet, oral hypoglycemic agents and insulin first when clinically needed
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — Insulin treatment in accordance to glucose values

SUMMARY:
Among adult patients diagnosed with type 2 diabetes, about 6% have autoantibodies directed against the insulin producing beta cells in the pancreas. These patients have a progressive beta cell destruction and most of them will be insulin dependent within 3-5 yrs. Patients with this latent autoimmune diabetes in adults (LADA) have a considerable remaining beta cell mass at diagnosis, and are suitable for evaluating new therapies for autoimmune diabetes Animal studies in diabetes prone mice have demonstrated potential positive effects of early insulin treatment, with a lower incidence of diabetes or a delay before diagnosis. The aim of this study was to investigate the effect of early insulin treatment of LADA patients, in respect to residual beta-cell function and metabolic control, compared to a group who were conventionally treated with diet and/or oral hypoglycaemic agents (OHA) and insulin not before it was clinically needed.

DETAILED DESCRIPTION:
All adult newly diagnosed diabetic patients in the certain areas are screened for pancreatic antibodies. Patients clinically classified as Type 2, not insulin requiring at diagnosis and positive for at least one autoantibody are eligible for inclusion. After randomisation to insulin treatment or diet and/or OHA, the patients are followed up with fasting C-peptide every third month. A glucagon test is performed, and stimulated C-peptide and HbA1c, + clinical data and body weight are recorded at baseline and after 12, 24 and 36 months. The final outcome of the study is C-peptide, and change in C-peptide compared to baseline level, and HbA1c, after 36 months.

ELIGIBILITY:
Inclusion Criteria:

* >18 yrs
* Positive for pancreatic autoantibodies

Exclusion Criteria:

* <18 yrs
* Significant concomitant diseases
* Not able to follow protocol

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 1995-02; Primary Completion 2002-04 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Glucagon stimulated C-peptide | 36 months after entering the study
  Glucagon stimulated C-peptide is measured at diagnosis and annually for three years. Basal values will be compared to values obtained after 36 months.